CLINICAL TRIAL: NCT01919619
Title: A Pilot Study of Lenalidomide Alternating With Ipilimumab Post Allogeneic and Autologous Stem Cell Transplantation
Brief Title: Lenalidomide and Ipilimumab After Stem Cell Transplant in Treating Patients With Hematologic or Lymphoid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0947; NCI-2013-02213 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012.0947; 2012-0947 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Hematopoietic and Lymphoid Cell Neoplasm; Leukemia; Lymphoma; Plasma Cell Myeloma; T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Lymphoma, T-Cell | interventions — Ipilimumab; CTLA-4 Antigen; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide and ipilimumab) (Experimental): Patients receive lenalidomide PO QD on days 1-21 of courses 1, 3, 5 and 7. Beginning 1-3 days after the last dose of lenalidomide patients receive one dose of ipilimumab IV over 90 minutes of courses 2, 4, 6 and 8. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Drug: Lenalidomide

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This pilot clinical trial studies the side effects of lenalidomide and ipilimumab after stem cell transplant in treating patients with hematologic or lymphoid malignancies. Biological therapies, such as lenalidomide, may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Immunotherapy with monoclonal antibodies, such as ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving lenalidomide with ipilimumab may be a better treatment for hematologic or lymphoid malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of lenalidomide in combination with ipilimumab in autologous and allogeneic stem cell transplantation.

SECONDARY OBJECTIVES:

I. Overall response rate. II. Overall survival, progression-free survival. III. Cumulative incidence of acute and chronic graft-versus-host disease (GVHD) with the competing risk of relapse in allogeneic transplant patients.

OUTLINE:

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21 of courses 1, 3, 5 and 7. Beginning 1-3 days after the last dose of lenalidomide patients receive one dose of ipilimumab intravenously (IV) over 90 minutes of courses 2, 4, 6 and 8. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 3, 6, 12, 24, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic or lymphoid malignancy
* Autologous patients can be included anytime within 6 months post-transplant, if they had no signs of progression and meet one of the following criteria: i. leukemia; ii. lymphoma (all types of B and T cell lymphoma); iii. multiple myeloma
* Allogeneic patients if: i. patients had engrafted donor cells (i.e., > 20% donor T-cell from peripheral blood [PB]/polymerase chain reaction [PCR]); and, ii. patients NOT in complete remission (CR) after their allogeneic transplant, and off tacrolimus and/or mycophenolate mofetil for at least 3 to 4 weeks with no signs of GVHD; or, iii. patients had evidence of relapse after their transplant who are off tacrolimus and/or mycophenolate mofetil or other immunosuppressants for GVHD for 3 to 4 weeks with no signs of GVHD (prednisone doses =< 10 mg are permitted as stated previously)
* No active infection
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets > 75 x 10^9/L
* Able to adhere to the study visit schedule and other protocol requirements
* Performance status: Eastern Cooperative Oncology Group (ECOG) 2 or less or Karnofsky of at least 60
* Cardiac ejection fraction (EF) >= 45% by 2-dimensional echocardiogram (2D-ECHO) within 3 months of study entry (or within 1 month if received chemotherapy within the past 3 months)
* Forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and diffusing capacity of the lung for carbon monoxide (DLCO) >= 40% within 3 months of study entry (or within 1 month if received chemotherapy within the past 3 months)
* Serum creatinine =< 1.6 mg/dL and creatinine clearance >= 30 ml/min; creatinine clearance will be calculated using the Cockcroft-Gault equation
* Serum glutamate pyruvate transaminase (SGPT), serum glutamic oxaloacetic transaminase (SGOT) less than 2 x the upper limit of normal range (unless related to Gilbert's disease or medications)
* Direct bilirubin < 1.6 (unless related to Gilbert's disease or medications)
* Patient or legally authorized representative able to sign informed consent
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to study entry

Exclusion Criteria:

* Immunotherapy or chemotherapy with approved or investigational anticancer therapeutics within 4 weeks of first dose
* Patients on alemtuzumab within 6 weeks prior to consenting
* Active congestive heart failure (New York Heart Association [NYHA] class III to IV), symptomatic ischemia or conduction abnormalities uncontrolled by conventional interventions; myocardial infarction within 6 months of study entry
* Deep vein thrombosis or pulmonary embolism within 3 months of study entry
* Pregnant or breast-feeding females; (lactating females must agree not to breast-feed while taking lenalidomide)
* Acute active infection requiring intravenous antibiotics, antiviral (except antiviral directed at hepatitis B), or antifungal agents within 14 days of first dose
* Known human immunodeficiency virus (HIV) seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen [Sag] or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed)
* Patients with other known malignancies within the past three years except: i. adequately treated basal or squamous cell skin cancer; ii. carcinoma in situ of the cervix; iii. prostate cancer with Gleason score < 6 with stable prostate-specific antigen (PSA) over the past three months; iv. breast cancer in situ with full surgical resection
* Significant neuropathy (grades 3 to 4 or grade 2 pain)
* Known hypersensitivity to thalidomide, lenalidomide or ipilimumab
* Active life-threatening autoimmune disease
* Active GVHD or recent GVHD and still on > 10 mg prednisone (or equivalent)
* Prior auto-immune disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa Khouri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Khouri IF, Fernandez Curbelo I, Turturro F, Jabbour EJ, Milton DR, Bassett RL Jr, Vence LM, Allison JP, Gulbis AM, Sharma P. Ipilimumab plus Lenalidomide after Allogeneic and Autologous Stem Cell Transplantation for Patients with Lymphoid Malignancies. Clin Cancer Res. 2018 Mar 1;24(5):1011-1018. doi: 10.1158/1078-0432.CCR-17-2777. Epub 2017 Dec 15. PMID 29246938
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered in MD Anderson Cancer Center
Groups:
- Autologous -Treatment (Lenalidomide and Ipilimumab); Allogeneic - Treatment (Lenalidomide and Ipilimumab): Patients receive lenalidomide PO QD on days 1-21 of courses 1, 3, 5 and 7. Beginning 1-3 days after the last dose of lenalidomide patients receive one dose of ipilimumab IV over 90 minutes of courses 2, 4, 6 and 8. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Ipilimumab: Given IV
  Lenalidomide: Given PO
Period: Overall Study
Arm/Group | Autologous -Treatment (Lenalidomide and Ipilimumab) | Allogeneic - Treatment (Lenalidomide and Ipilimumab)
Started | 28 | 13
Completed | 27 | 12
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous -Treatment (Lenalidomide and Ipilimumab) | Allogeneic - Treatment (Lenalidomide and Ipilimumab) | Total
Number analyzed (Participants) | 28 | 13 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 10 | 33
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 19 | 7 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 25 | 12 | 37
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 13 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experienced Severe Toxicity From Lenalidomide and Ipilimumab Post Transplant
Description: Any grade 4 hematological toxicity or grade 3-5 organ toxicity 30 days following the last dose of study drug.
Time Frame: Up to 30 days following the last dose of study drugs
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous -Treatment (Lenalidomide and Ipilimumab) | Allogeneic - Treatment (Lenalidomide and Ipilimumab)
Number analyzed (Participants) | 28 | 13
Participants | 10 | 2

2. Secondary Outcome: Number of Participants Achieved Complete Remission
Description: CR is defined as a complete resolution of all target lesions by CT scans with complete normalization of FDG-PET uptake in all areas, and bone marrow biopsy negativity.
Time Frame: Up to 30 days following the last dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous -Treatment (Lenalidomide and Ipilimumab) | Allogeneic - Treatment (Lenalidomide and Ipilimumab)
Number analyzed (Participants) | 28 | 13
Participants | 22 | 5

3. Secondary Outcome: Progression-free Survival
Description: Number of participants that are alive and disease free 36 months long post transplant
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous -Treatment (Lenalidomide and Ipilimumab) | Allogeneic - Treatment (Lenalidomide and Ipilimumab)
Number analyzed (Participants) | 28 | 13
Participants | 18 | 4

ADVERSE EVENTS:
Time Frame: up to 36 months
Arm/Group | Autologous -Treatment (Lenalidomide and Ipilimumab) | Allogeneic - Treatment (Lenalidomide and Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 7/28 | 5/13
Serious Adverse Events (participants affected / at risk) | 10/28 | 2/13
Other Adverse Events (participants affected / at risk) | 25/28 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous -Treatment (Lenalidomide and Ipilimumab) (N=28) | Allogeneic - Treatment (Lenalidomide and Ipilimumab) (N=13)
Low granulocyte (Blood and lymphatic system disorders) | 10 (10) | 2 (2)
Low platelet (Investigations) | 0 (0) | 1 (1)
Viral (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous -Treatment (Lenalidomide and Ipilimumab) (N=28) | Allogeneic - Treatment (Lenalidomide and Ipilimumab) (N=13)
Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
ALK increased (Investigations) | 12 (12) | 2 (2)
AL OTH (General disorders) | 0 (0) | 1 (1)
ALT increased (Investigations) | 13 (13) | 7 (7)
Anemia (Investigations) | 22 (22) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
AST increased (Investigations) | 13 (13) | 6 (6)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Bacterial (Infections and infestations) | 1 (1) | 2 (2)
Blurred vision (Eye disorders) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Creatinine increased (Investigations) | 7 (7) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (15) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dysrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Edema (General disorders) | 2 (2) | 0 (0)
EN OTH (Endocrine disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 9 (9) | 4 (4)
Fever (General disorders) | 3 (3) | 0 (0)
Flu like syndrome (General disorders) | 5 (5) | 5 (5)
Fluid overload (General disorders) | 0 (0) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GI OTH (Gastrointestinal disorders) | 1 (1) | 3 (3)
GU OTH (Renal and urinary disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypertension (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
IN FEC (Infections and infestations) | 3 (3) | 3 (3)
LDH increased (Investigations) | 6 (6) | 0 (0)
Low granulocyte (Blood and lymphatic system disorders) | 22 (48) | 13 (13)
Low platelet (Investigations) | 25 (25) | 13 (13)
Lymphocytosis (Investigations) | 1 (1) | 1 (1)
MT OTH (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (4)
NE OTH (Nervous system disorders) | 4 (4) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Other (General disorders) | 10 (10) | 3 (3)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PU OTH (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 12 (12) | 4 (4)
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
T bilirubin increased (Investigations) | 4 (4) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
Viral (Infections and infestations) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Wbc decreased (Investigations) | 20 (38) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT01919619/Prot_SAP_000.pdf